CLINICAL TRIAL: NCT04150822
Title: Hereditary Hemorrhagic Telangiectasia (HHT) Research Outcomes Registry
Brief Title: CHORUS - Comprehensive HHT Outcomes Registry of the United States (Formerly OUR HHT Registry)
Status: Active, not recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Cure HHT (Other); Dartmouth College (Other)
Responsible Party: Sponsor
Other Study IDs: OURHHT
Record Dates: First submitted 2019-09-18; First posted 2019-11-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; HHT; Arteriovenous Malformation of Brain
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Arteriovenous Malformations | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Registry and Saliva sample — Non-interventional registry with saliva sample collected for DNA analysis

SUMMARY:
The goal of this study is to better understand HHT, the symptoms and complications it causes ("outcomes") and how the disease impacts people's lives. The investigators are aiming to recruit and gather information together in the Registry from 1,000 HHT patients from four HHT Centres of Excellence in North America. The Investigators will collect long-term information about the people in the Registry, allowing the investigators to understand how the disease changes over time, and what factors can influence those changes. Ultimately, this should help improve treatments for the disease.

DETAILED DESCRIPTION:
Background and Rationale HHT has an estimated prevalence of 1 in 5000, affecting children and adults, in multiple organs. The disease is characterized by the presence of vascular malformations (VMs), including arteriovenous malformations (AVMs) of the lung, liver, brain, spinal cord and smaller mucosal lesions (telangiectasia) of the nose, mouth and GI tract. These lesions lead to acute and chronic bleeding, stroke, heart failure and death. Treatments are currently mostly limited to managing complications, while approximately 90% of adults have ongoing symptoms, despite best surgical and medical therapies. With recent drug development related to angiogenesis, there is hope for effective novel therapies. Investigators, experts, the International HHT Guidelines, Pharma representatives, the CDC and HHT patient advocates (curehht.org) all agree that there is an urgent need for natural history data in this disease, with characterization of clinical outcomes, to allow patients to benefit from the explosion of drug development in the field.

As of August 27, 2023, the OUR HHT Registry has transitioned to the CHORUS platform (Studytrax) for ongoing data collection. Only select CHORUS-funded sites are currently enrolling. The Toronto site has completed enrollment but remains active with REB approval.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with HHT by the Curacao criteria (either 3+ clinical diagnostic criteria or genetic diagnosis).
* Capable of giving informed consent in person or via a substitute decision maker
* >18 years

Exclusion Criteria:

* Participants unable to give informed consent either in person or with a substitute decision maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Hereditary Hemorrhagic Telangiectasia (HHT), living in North America
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Prospective and longitudinal characterization of major outcomes of HHT in a cohort of HHT patients, from Centers of Excellence in North America. | 10 Years
  Comprehensive baseline clinical, demographic and lifestyle data will be collected and entered into the recruitment-ready newly developed OUR HHT Registry.
The longitudinal characterization of major outcomes of HHT in the North American cohort | 10 Years
  Annual outcome data will be collected and entered into the recruitment-ready newly developed OUR HHT Registry.

SECONDARY OUTCOMES:
Characterizing the determinants of HHT by prospectively and longitudinally measuring the rates of clinical outcome of HHT | 10 Years
  The rates of severe complications of HHT will be measured and their determinants characterized.
Epistaxis which affects 90% of adults with HHT, will be characterized by measuring the rates of clinical outcome. | 10 Years
  The characteristics and determinants of epistaxis will be studied.
The prospective development of organ VMs in HHT patients | 10 Years
  Development of new VMs/growth of VMs and its determinants will be measured.
The rates of venous thromboembolism (VTE) in HHT patients | 10 Years
  The rates and determinants of venous thromboembolism in HHT patients will be measured prospectively.
A DNA repository of HHT subjects will be created as a resource for future genetic, pharmacogenetics and targeted therapy studies. | 10 Years
  Saliva samples of all recruited subjects will collected to create a DNA repository

OTHER OUTCOMES:
Participant entered data | 10 Years
  Data collection from participant relating symptoms and knowledge of HHT

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Faughnan, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided